CLINICAL TRIAL: NCT07237854
Title: Effect of Continuous Versus High-intensity Interval Aerobic Training on the Muscular Vascular Adaptation
Brief Title: Effect of Training Intensity on Microvascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Emilie Maufroy, Research Scientist, Reasearch Unit in Rehabilitation Sciences, Université Libre de Bruxelles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ULB
Record Dates: First submitted 2022-09-26; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Vascular Remodeling; Sedentary Behavior; Hemodynamic Rebound
Keywords: Microcirculation; Hemodynamic Instability; Microvascular Density; Quadriceps Muscle; Endurance Training; High-Intensity Interval Training
MeSH Terms: conditions — Vascular Remodeling; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A parallel group randomised controlled trial will be used to determine the superiority of high-intensity interval training versus continuous training on the improvement of quadricpes microvascular function.
Masking Description: Participants and the researcher will know the group allocation and therfore cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Continuous Training (MICT): 34 min at 65% maximal heart rate (Experimental): Participants performed a 3-minute warm-up at 50% of their maximal heart rate (HRmax), as determined during baseline cardiopulmonary exercise testing (ergospirometry), followed by 40 minutes of continuous cycling at 65% of their VO₂max. Sessions were conducted three times per week for a total duration of 8 weeks.
  Interventions: Procedure: Percutaneous muscle biopsies of the vastus lateralis (quadriceps); Other: Measurement of the maximal oxygen uptake (VO2max); Other: Non-Invasive Cardiac Output Measurement (Innocor)
- High-Intensity Interval Training (HIIT): 2x2 min at 65% and 90% of maximal heart rate (Experimental): Participants performed a 3-minute warm-up at 50% of their maximal heart rate (HRmax), as determined during baseline cardiopulmonary exercise testing (ergospirometry). The main training protocol consisted of alternating 2-minute cycling bouts: 2 minutes at 65% HRmax followed by 2 minutes at 90% HRmax, repeated continuously for a total of 28 minutes. Sessions were conducted three times per week over an 8-week period.
  Interventions: Procedure: Percutaneous muscle biopsies of the vastus lateralis (quadriceps); Other: Measurement of the maximal oxygen uptake (VO2max); Other: Non-Invasive Cardiac Output Measurement (Innocor)

INTERVENTIONS:
Procedure: Percutaneous muscle biopsies of the vastus lateralis (quadriceps) — Percutaneous muscle biopsies of the vastus lateralis (quadriceps) were performed under local anesthesia. Samples were collected at baseline and/or post-intervention to assess microvascular structure, fiber composition, and molecular adaptations to aerobic training.
Other: Measurement of the maximal oxygen uptake (VO2max) — Cardiopulmonary Exercise Testing (CPET) Maximal oxygen consumption (VO₂max) was assessed using an incremental stepwise protocol on a cycle ergometer. Participants performed the test at baseline and after the 8-week training intervention. Respiratory gas exchange was continuously measured using a COSMED K5 portable metabolic system, which provided breath-by-breath analysis of oxygen uptake (VO₂), carbon dioxide production (VCO₂), and ventilation parameters. The test was terminated upon volitional exhaustion or when predefined criteria for VO₂max plateau were met.
Other: Non-Invasive Cardiac Output Measurement (Innocor) — Maximal cardiac output was assessed at peak exercise intensity during cardiopulmonary exercise testing (CPET) using the Innocor device. This system employs the inert gas rebreathing technique, which involves the controlled inhalation of a gas mixture containing nitrous oxide (N₂O) and sulfur hexafluoride (SF₆). By analyzing the washout kinetics of these gases during rebreathing, the device estimates pulmonary blood flow, which is then used to calculate cardiac output non-invasively. Measurements were performed at the maximal workload reached during the incremental cycling test.

SUMMARY:
The aim of this trial is to investigate the effect of aerobic training intensity on muscle vascular function: continuous versus interval.

DETAILED DESCRIPTION:
This trial will compare the hemodynamic effects of aerobic training on muscle microvascular function between participants randomly assigned to one of two groups: a continuous training group and an high-intensity interval training group.

All data concerning the primary and secondary outcomes will be obtained at the start and repeated at the end of 8 weeks aerobic training.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female or male between 18 and 45 years
* Be sedentary
* Able to cycle
* Able to provide written informed consent

Exclusion Criteria:

* Have a pathology that may impact vascular function as :

  * cardiac pathology
  * pneumological pathology
  * metabolic pathology
* Smoke

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percutaneous muscle biopsies of the vastus lateralis | At baseline and after completion of the 8-week intervention
  Muscle tissue samples obtained from the vastus lateralis were processed using optical clearing and immunohistochemical staining techniques to visualize the microvascular network. Confocal microscopy was employed to acquire high-resolution three-dimensional images of arterioles, capillaries, and venules. Quantitative assessments included:
  1. Internal diameter measurements, based on endothelial cell boundaries (intima layer)
  2. External diameter measurements, based on smooth muscle cells and pericytes (media layer)
  3. Capillary density, determined by counting the number of capillaries per sample volume

SECONDARY OUTCOMES:
Cardiopulmonary Exercise Testing (CPET) | At baseline and after completion of the 8-week intervention
  VO₂max was determined using a graded, incremental exercise test performed on a cycle ergometer until volitional exhaustion. Throughout the test, respiratory gases were continuously measured using a metabolic cart (e.g., COSMED K5), which provided breath-by-breath analysis.
  The following parameters were recorded :
  1. VO₂ (oxygen uptake) in mL/min
  2. VCO₂ (carbon dioxide production) in mL/min
  3. Minute ventilation (VE) in L/min
Maximal Cardiac Output Measurement Using Inert Gas Rebreathing (Innocor) | At baseline and after completion of the 8-week intervention
  Innocor is a medical device that estimates cardiac output using the inert gas rebreathing technique, a validated non-invasive method. During the procedure, the participant inhales a gas mixture containing nitrous oxide (N₂O) and sulfur hexafluoride (SF₆) through a closed circuit. These inert gases are absorbed and eliminated at rates proportional to pulmonary blood flow. By analyzing the washout kinetics of these gases during a brief rebreathing period, Innocor calculates pulmonary blood flow, which is then used to estimate cardiac output. This measurement is typically performed at rest or at peak exercise intensity, such as during the final stage of a cardiopulmonary exercise test (CPET).
  The system provides real-time data on:
  1. Cardiac output (L/min)
  2. Stroke volume (ml/min)
  3. Heart rate (bpm)
  4. Pulmonary blood flow (L/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Université Libre de Bruxelles, Faculté des Sciences de la motricité, Laboratoire de kinésithérapie, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: No